CLINICAL TRIAL: NCT02093910
Title: Phase 2 Study of Concurrent Monosialotetrahexosylganglioside in the Prophylactic Treatment of Bortezomib-induced Peripheral Neuropathy in Patients of Multiple Myeloma
Brief Title: Efficacy of Monosialotetrahexosylganglioside in the Prophylactic Treatment of Bortezomib-induced Peripheral Neuropathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xia Zhongjun, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GM1
Record Dates: First submitted 2014-03-13; First posted 2014-03-21 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; peripheral neuropathy; prophylaxis
MeSH Terms: conditions — Multiple Myeloma; Peripheral Nervous System Diseases | interventions — G(M1) Ganglioside; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Monosialotetrahexosylganglioside (Experimental): each patient in this arm received velcade+dexamethasone (VD) regimen（bortezomib,1.3mg/㎡，subcutaneously injection，d1,8,15,22；dexamethasone,20mg d1-2, 8-9,15-16,22-23）every 4 weeks; and monosialotetrahexosylganglioside was used at the dosage of 100mg/d intravenously at d1-2,8-9,15-16,22-23 every cycle.
  Interventions: Drug: Monosialotetrahexosylganglioside

INTERVENTIONS:
Drug: Monosialotetrahexosylganglioside
  Other Names: bortezomib; dexamethasone

SUMMARY:
Bortezomib was an important drug in the treatment of multiple myeloma (MM),and peripheral neuropathy (PN) is a significant dose-limiting toxicity of bortezomib that typically occurs within the first courses of bortezomib, reaches a plateau at cycle 5. Up to now, no effective prophylaxis have been developed for PN. Monosialotetrahexosylganglioside, a nerve-protecting drug,was often used to promote growth of nerve, and function restoration of damaged nerve.Thus,the investigators hypothesized that combination of Monosialotetrahexosylganglioside and bortezomib can reduce the incidence rate of peripheral neuropathy (PN) and promote the relief of peripheral neuropathy (PN) in multiple myeloma (MM) patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of multiple myeloma;
* Age:18-80 years;
* Eastern Cooperative Oncology Group (ECOG) status 0-3,
* Estimated survival time > 3 months;
* Acceptable liver function (bilirubin<2.5×ULN, Alanine transaminase (ALT) or Aspartate Aminotransferase (AST)<2.5×ULN),
* No history of other malignancies;
* No previous treatments including chemotherapy, radiotherapy, targeted therapy or stem cell transplantation;
* No other serious diseases which conflict with the treatment in the present trial;
* No concurrent treatments that conflict with the treatments in the present trial;
* Voluntary participation and signed the informed consent.

Exclusion Criteria:

* The patients had the conditions below: clinically significant ventricular tachycardia (VT), atrial fibrillation (AF), heart block, myocardial infarction (MI), congestive heart failure (CHF), symptomatic coronary artery heart disease requiring medication;
* The patients participated in other clinical trials within the 30 days before enrollment or who are participating in other clinical studies;
* The patients with neuropathy;
* The patients with mentally ill / unable to obtain informed consent;
* The patients with drug addiction, alcohol abuse which affects the long-term evaluation of test results;
* The patients in pregnancy, lactation and women of childbearing age who do not want to take contraceptive measures subjects;
* The patients with a history of allergy to test drug;
* The patients not suitable to participate in the investigator judged by researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
overall incidence rate of peripheral neuropathy (PN) | up to 6 months
  the grade of peripheral neuropathy (PN) was recorded according to Common Terminology Criteria for Adverse Events (CTCAE) v3.0.

SECONDARY OUTCOMES:
duration of peripheral neuropathy (PN) | up to 1 year (about 6 months after the completion of treatment)
  the duration of peripheral neuropathy means the time from the onset time of peripheral neuropathy (PN) to the relief time of PN
complete rate (CR) rate | up to 6 months
  The criteria for CR was according to International Myeloma Working Group Uniform Response Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-jun Xia, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center; State Key Laboratory of Oncology in South China,, Guangzhou, Guangdong, China